CLINICAL TRIAL: NCT06511128
Title: Evaluation of Anesthesia Depth Using 4-channel EEG in Patients Undergoing Drug-induced Sleep Endoscopy (DISE) With Two Different Sedation Methods.
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: TABED 1-24-36
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Seeing the Benefits of Using 4 Channel EEG During the DISE Procedure With Sedation
Keywords: 4 channel EEG; sedasyon; uyku endoskopisi; propofol; dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — biospecimens are not used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group created with dexmedetomidine sedation: infusion will be started at a dose of 0.2-0.7 mcg/kg/h after a loading dose of 1 mg midazolam, 50 mcg fentanyl followed by 1 mcg/kg dexmetedomidine.
- group created with propofol sedation: After 1 mg midazolam and 50 mcg fentanyl are given, propofol infusion will be started at a dose of 50-100 mcg/kg/min, following an initial dose of 0,5 mg/kg

SUMMARY:
You will undergo a drug-induced sleep endoscopy procedure. The drugs we use to create routine sedation will be used as medication. During the procedure, your pulse, blood pressure, respiratory rate, blood oxygen level, and alertness will be monitored. Your values will be closely monitored and recorded before, during and after the procedure.

Our study is a study that will not require any changes in the drug-induced sleep endoscopy (DISE) procedure and treatment plan you will undergo. During drug-induced sleep endoscopy (DISE), your measurement values, which we follow in every patient, will be recorded. An adhesive tape will be attached to your forehead area, especially to determine your sleep depth. It will be removed at the end of the procedure.

DETAILED DESCRIPTION:
Volunteer patients between the ages of 18-65, both genders and ASA (American Society of Anesthesiology) I-II risk scores, who will undergo DISE with sedation after routine preoperative evaluation under elective conditions, will be included in the study.All patients participating in the study will be explained about the study and possible risks and informed consent will be obtained from the patients.

Exclusion criteria for the study: Patient unwillingness, being younger than 18 years of age, being older than 65 years of age, patients with ASA score greater than II, pregnant women, drug addicts, alcohol addicts, patients with congestive heart failure, need for intubation, patients receiving oxygen therapy at home, Patients with chronic analgesic use, patients known to be allergic to the anesthetic drugs used, patients with psychiatric disorders.

The patient age, weight, BMI, AHI index if any, existing chronic diseases, medications used, whether or not CPAP has been used at home for how many years, duration of the procedure, amount of medications used, whether the airway is intervened or not, hemodynamic(systolic arterial pressure, diastolic arterial pressure, average parameters (e.g. arterial pressure, heart rate, oxygen saturation) will be recorded throughout the procedure.

At the end of the procedure, the patient will be taken to the recovery unit and will be evaluated according to Aldrete criteria and if there is no problem, patient will be sent to the service.The patient's wake-up time, recovery time, and possible complications during recovery will be noted and treatment will be planned.

All patients entering the operating room will receive ASA monitoring (non-invasive arterial blood pressure, ECG, oxygen saturation) followed by 4-channel EEG monitoring and baseline values will be noted.After a 4lt/min nasal oxygen cannula is placed, 1 mg midazolam and 50 mcg fentanyl will be given to group I, and then propofol infusion will be started at a dose of 50-100 mcg/kg/min, following an initial dose of 1mg/kg.In group II, infusion will be started at a dose of 0.2-0.7 mcg/kg/h after a loading dose of 1 mg midazolam, 50 mcg fentanyl followed by 1 mcg/kg dexmetedomidine.Anesthesia depth dose adjustment will be made according to the 60-70 PSI value range in the 4-channel EEG. The time to reach the adequate processing level will be recorded.Patients who have reached the target depth of sedation but have hypertension will be given an additional 0.1 mg of glyceryl trinitrate.Decreases of 25% from baseline blood pressure will be considered hypotension and will be treated with fluid boluses and/or followed by IV ephedrine.In the event of apnea or desaturation, airway management techniques such as patient stimulation, increased oxygen supplementation, chin lift, chin thrust maneuver will be applied and noted.

If the pulse rate drops below 50 bpm, treatment with IV 0.5 mg atropine will be considered. While the patient is being sent to the ward, the patient will be asked whether he or she has had a dream, and if so, its content will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patients of both genders and ASA (American Society of Anesthesiology) I-II risk scores, between the ages of 18-65, who will undergo DISE with sedation.

Exclusion Criteria:

* Patient unwillingness, being younger than 18 years of age, being older than 65 years of age, patients with ASA score greater than II, pregnant women, drug addicts, alcohol addicts, patients with congestive heart failure, need for intubation, patients receiving oxygen therapy at home, Patients with chronic analgesic use, patients known to be allergic to the anesthetic drugs used, patients with psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA I-II patients between the ages of 18-65 who will undergo sleep endoscopy under sedation in the operating room of Ankara City Hospital Ear Nose and Throat Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Determination of sedation range in 4-channel EEG | from March 2024 to December 2024
  Evaluation of sedation depth using 4-channel EEG in drug-induced sleep endoscopy (DISE)"

SECONDARY OUTCOMES:
Evaluating the effectiveness of different sedation techniques,Snoring situation in the shortest time and effectively,Intraoperative drug consumption,Hemodynamic changes | from March 2024 to December 2024
  Evaluating the effectiveness of different sedation techniques,Snoring situation in the shortest time and effectively,Intraoperative drug consumption,Hemodynamic changes

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi e Erkılıç, doc doctor, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No